CLINICAL TRIAL: NCT03796858
Title: Phase 3b, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Guselkumab Administered Subcutaneously in Participants With Active Psoriatic Arthritis and an Inadequate Response to Anti-Tumor Necrosis Factor Alpha (Anti-TNFα) Therapy
Brief Title: A Study of Guselkumab in Participants With Active Psoriatic Arthritis and an Inadequate Response to Anti-Tumor Necrosis Factor Alpha (Anti-TNF Alpha) Therapy
Acronym: COSMOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108573; 2018-003214-41 (EudraCT Number); CNTO1959PSA3003 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2019-01-07; First posted 2019-01-08 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Guselkumab (Experimental): Participants will receive guselkumab 100 milligram (mg) Subcutaneous (SC) injection at Weeks 0, 4, 12, 20, 28, 36, and 44 and placebo SC at Week 24 to maintain the blind. At Week 16, Participants who meet the early escape criteria will receive placebo at Week 16 and guselkumab at Week 20, then guselkumab every 8 weeks (q8w).
  Interventions: Drug: Guselkumab 100 mg; Drug: Placebo
- Group 2: Placebo followed by Guselkumab (Experimental): Participants will receive placebo SC injection at Weeks 0, 4, 12, and 20, and will crossover to receive guselkumab 100 mg SC injection at Weeks 24, 28, 36, and 44. At Week 16, Participants who meet the early escape criteria will receive guselkumab at Weeks 16 and 20, then guselkumab q8w.
  Interventions: Drug: Guselkumab 100 mg; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab 100 mg — Participants will receive guselkumab 100mg as SC injection.
  Other Names: CNTO 1959
Drug: Placebo — Participants will receive placebo as SC injection.

SUMMARY:
The purpose of this study is to evaluate guselkumab efficacy versus placebo in participants with active psoriatic arthritis (PsA) and an inadequate response to Anti-Tumor Necrosis Factor Alpha (TNF-alpha) therapy by assessing the reduction in signs and symptoms of joint disease.

DETAILED DESCRIPTION:
Psoriatic arthritis is a multi-faceted disease that impacts the joints, soft tissues, and skin, all of which not only results in functional disability and impaired quality of life, but participants with this disease also have increased mortality. Guselkumab is a monoclonal antibody that binds to human interleukin 23 (IL-23) and inhibits IL-23 specific intracellular signaling and subsequent activation and cytokine production. Investigation of guselkumab in this Phase 3b PsA clinical study is supported by the favorable efficacy and safety results from Phase 2 study of guselkumab in PsA and Phase 2 and Phase 3 studies in psoriasis including the subset of participants with PsA. The primary hypothesis is that guselkumab 100 milligram (mg) at Weeks 0, 4, and every 8 weeks (q8w) thereafter is superior to placebo which will be assessed by the proportion of participants achieving an American College of Rheumatology (ACR 20) response at Week 24. The study includes 2 periods: A 24-week double-blind, placebo-controlled period for the primary analysis of the efficacy and safety of guselkumab, compared with placebo and a 32-week active-treatment and safety follow-up period for additional analysis of the efficacy and safety of guselkumab. Safety will be monitored throughout the study (Up to Week 56).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of psoriatic arthritis (PsA) for at least 6 months before the first administration of study intervention and meet classification criteria for Psoriatic Arthritis (CASPAR) at screening
* Have active PsA as defined by at least 3 swollen joints and at least 3 tender joints at screening and at baseline
* Have at least 1 of the PsA subsets: distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Have an inadequate response to anti-TNF alpha therapy, defined as presence of active PsA despite previous treatment with either 1 or 2 anti-TNF alpha agents and either of the following: a) Lack of benefit of an anti-TNF alpha therapy, as documented in the participant history by the treating physician, after at least 12 weeks of etanercept, adalimumab, golimumab, or certolizumab pegol therapy (or biosimilars) and/or at least a 14-week dosage regimen (i.e., at least 4 doses) of infliximab (or biosimilars). Documented lack of benefit may include inadequate improvement in joint counts, skin response, physical function, or disease activity, b) Intolerance to an anti-TNF alpha therapy, as documented in the patient history by the treating physician, to etanercept, adalimumab, golimumab, certolizumab pegol, or infliximab (or biosimilars, if available)
* Be willing to refrain from the use of complementary therapies for PsA or psoriasis including ayurvedic medicine, traditional Taiwanese, Korean, or Chinese medications and acupuncture within 2 weeks before the first study intervention administration and through Week 48

Exclusion Criteria:

* Has other inflammatory diseases that might confound the evaluations of benefit of guselkumab therapy, including but not limited to rheumatoid arthritis (RA), axial spondyloarthritis (this does not include a primary diagnosis of PsA with spondylitis), systemic lupus erythematosus, or Lyme disease
* Has ever received more than 2 different anti-TNF alpha agents
* Has previously received any biologic treatment (other than anti-TNF Alpha agents), including, but not limited to ustekinumab, abatacept, secukinumab, tildrakizumab, ixekizumab, brodalumab, risankizumab, or other investigative biologic treatment
* Has previously received tofacitinib, baricitinib, filgotinib, peficitinib (ASP015K), decernotinib (VX 509), or any other a Janus kinase (JAK) inhibitor
* Has previously received any systemic immunosuppressants (for example, azathioprine, cyclosporine, 6 thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus) within 4 weeks of the first administration of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve an American College of Rheumatology (ACR) 20 Response at Week 24 | Week 24
  The ACR 20 Response is defined as greater than or equal to (>=) 20 percent (%) improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=20 percent improvement in 3 of following 5 assessments: participant's assessment of pain using Visual Analog Scale (VAS; 0-10 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), participant's global assessment of disease activity by using VAS (scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and C-reactive protein (CRP).

SECONDARY OUTCOMES:
Change from Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24 | Baseline, Week 24
  The HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping and activities of daily living). Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area). Overall score is computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Percentage of Participants who Achieve an ACR 50 Response at Week 24 | Week 24
  The ACR 50 Response is defined as greater than or equal to (>=) 50 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=50 percent improvement in 3 of following 5 assessments: participant's assessment of pain using Visual Analog Scale (VAS; 0-10 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), participant's global assessment of disease activity by using VAS (scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and C-reactive protein (CRP).
Change from Baseline in 36-Item Short form Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 24 | Baseline, Week 24
  The SF-36 is a generic health survey with 36 items that measure functional health and well-being from the participant's perspective. The survey is summarized into 8 dimensions/scales: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH). The physical component summary measure is derived from 4 of the 8 health dimensions (aggregate of PF, RP, BP, and GH scales). The minimum score is 0 and the maximum score is 100. A higher score indicates a better health state.
Percentage of Participants who Achieve Psoriatic Area and Severity Index (PASI) 100 Response at Week 24 Among Participants with >=3% body Surface area Psoriatic Involvement and an Investigator's Global Assessment (IGA) Score of >=2 (Mild) at Baseline | Week 24
  PASI 100 response is defined as 100% improvement in PASI score from baseline (PASI score of 0). The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI scoring system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A higher score indicates more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (117):
- Belgium (4):
  - CHU Saint Pierre BXL, Brussels
  - Reuma Clinic, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Bulgaria (7):
  - Diagnostic - Consulting Center II-Pleven, Pleven
  - Medical Center Medconsult-Pleven, Pleven
  - Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - Multiprofile Hosptal for Active Treatment Eurohospital Plovdiv, Plovdiv
  - Medical Center Teodora, Rousse
  - Diagnostic Consulting Center No 17, Sofia
  - Military Medical Academy, Sofia
- France (8):
  - Hopital Pellegrin Tripode - CHU de Bordeaux, Bordeaux
  - CHU Lapeyronie, Montpellier
  - Centre Hospitalier Regional d'Orleans (CHRO) - Hopital La Source, Orléans
  - Hopital Lariboisiere, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - Hopital Cochin, Paris
  - Centre Hospitalier Universitaire de Toulouse - Hopital Purpan, Toulouse
  - CHU Trousseau - Service de Rhumatologie, Tours
- Germany (6):
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Hamburger Rheuma Forschungszentrum II, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Rheumazentrum Ruhrgebiet, Herne
  - Rheumatologische Schwerpunktpraxis, Rendsburg
  - Krankenhaus St. Josef, Wuppertal
- 424 Military Hospital of Thessaloniki, Thessaloniki, Greece
- Hungary (6):
  - Betegapolo Irgalmas Rend Budai Irgalmasrendi Korhaz, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktatokorhaz, Székesfehérvár
  - MAV Korhaz es Rendelointezet, Szolnok
  - Vital Medical Center Orvosi es Fogaszati Kozpont, Veszprém
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Policlinico Tor Vergata, Roma
  - Complesso Integrato Columbus, Rome
  - Humanitas Hospital, Rozzano (MI)
- Poland (8):
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Bydgoszcz
  - Centrum Kliniczno Badawcze, Elblag
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - NZOZ Lecznica MAK MED S C, Nadarzyn
  - Medycyna Kliniczna, Warsaw
  - Mazowieckie Centrum Reumatologii i Osteoporozy, Warsaw
  - WroMedica I Bielicka A Strzalkowska s c, Wroclaw
- Portugal (7):
  - Uls Almada Seixal - Hosp. Garcia de Orta, Almada
  - Uls Regiao Aveiro - Hosp. Infante D. Pedro, Aveiro
  - Uls Braga - Hosp. Braga, Braga
  - Ipr Inst Port de Reumatologia, Lisbon
  - Uls Lisboa Ocidental - Hosp. Egas Moniz, Lisbon
  - Uls Santa Maria - Hosp. Santa Maria, Lisbon
  - Ulsam - Hosp. Conde de Bertiandos, Ponte de Lima
- Russia (19):
  - Chelyabinck Regional Clinical Hospital, Chelyabinsk
  - Kemerovo State Medical University, Kemerovo
  - Medical Centre Maximum Health, Kemerovo
  - Family polyclinic #4, Korolyov
  - Krasnodar Clinical Dermatovenerologic Dispensary, Krasnodar
  - Krasnoyarsk State Medical University, Krasnoyarsk
  - Orenburg State Medical Academy, Orenburg
  - Rostov Regional Clinical Dermatovenerological Dispensary, Rostov
  - Ryazan Regional Clinical Dermatovenerological Dispensary, Ryazan
  - Leningrad region clinical hospital, Saint Petersburg
  - Samara Regional Clinical Hospital Named After V.D.Seredavin, Samara
  - Sararov Regional Clinical Hospital, Saratov
  - Smolensk regional hospital on Smolensk railway station, Smolensk
  - Tula Regional Clinical Dermatovenerological Dispensary, Tula
  - Republican Clinical Hospital - G.G. Kuvatov, Ufa
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - Regional Clinical Hospital, Veliky Novgorod
  - Clinical Emergency Hospital n.a. N.V. Solovyev, Yaroslavl
  - Clinical Hospital #3, Yaroslavl
- Spain (15):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp. Univ. Germans Trias I Pujol, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. de Getafe, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. Infanta Luisa, Seville
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Ntra. Sra. de Valme, Seville
  - Hosp. Do Meixoeiro, Vigo
- Ukraine (15):
  - Communal Noncommercial Enterprise Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - Ivano-Frankivsk National Medical University, Ivano-Frankivsk City Clinical Hospital, Ivano-Frankivsk
  - City Multifield Hospital #18, Mechnikov Institute of Microbiology and Immunology of NAMS, Kharkiv
  - Municipal non-commercial enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - Khmelnitckiy regional hospital, Khmelnytsky
  - Kyiv City Clinical Hospital #3, National Medical University, Kyiv
  - Medical Center 'Consylium Medical', Kyiv
  - Kyiv Railway Station Clinical Hospital #2, Kyiv
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - ME Poltava Regional Clinical Hospital named after M.V. Sklifosovsky of Poltava Regional Consuil, Poltava
  - Municipal Institution of Sumy Regional Council Sumy Regional Clinical Hospital, Sumy
  - Municipal Non-commercial Enterprise Ternopil University Hospital of Ternopil Regional Council, Ternopil
  - Medical Center LTD Health Clinic Department of Cardiology and Rheumatology, Vinnytsia
  - VNMUn.af.Pyrogova,CNE Vinnytsia Regional Clinical Hospital n.af.Pyrogova Vinnytsia Regional Council, Vinnytsia
  - Municipal institution Central Clinical Hospital #1 Zhytomir, Zhytomyr
- United Kingdom (10):
  - Royal National Hospital for Rheumatic Diseases, Bath
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cannock Chase Hospital, Cannock
  - Chapel Allerton Hospital, Leeds
  - Barts Health NHS Trust Whipps Cross University Hospital NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust - Rheumatoid Arthritis (RA) Clinic, London
  - North Tyneside General Hospital, Newcastle
  - Peterborough City Hospital, Peterborough
  - Haywood Hospital, Stoke-on-Trent
  - Torbay Hospital-Devon, Torquay

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials\transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Gossec L, Baraliakos X, Galloway J, Oke V, Sfikakis P, Rampakakis E, Sharaf M, Lavie F, McInnes IB. Guselkumab Improves Patient-Reported Outcomes Among Participants with Psoriatic Arthritis and Inadequate Response to Tumor Necrosis Factor Inhibitors in the COSMOS Study. Rheumatol Ther. 2026 Jan 23. doi: 10.1007/s40744-025-00821-2. Online ahead of print. PMID 41575731
- [Derived] Gladman DD, Eder L, Selmi C, Mease PJ, Ogdie A, Lozenski K, Adamson E, Sharaf M, Rampakakis E, Pina Vegas L, Coates LC. Influence of Biological Sex on Participant Characteristics, Guselkumab Efficacy and Radiographic Progression in Active Psoriatic Arthritis: Post Hoc Analysis of Three Randomized Trials. Rheumatol Ther. 2025 Dec 15. doi: 10.1007/s40744-025-00812-3. Online ahead of print. PMID 41396391
- [Derived] Warren RB, McInnes IB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, Mease PJ. Comparative Effectiveness of Bimekizumab and Guselkumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):829-839. doi: 10.1007/s40744-024-00659-0. Epub 2024 Mar 15. PMID 38488975
- [Derived] Strober B, Coates LC, Lebwohl MG, Deodhar A, Leibowitz E, Rowland K, Kollmeier AP, Miller M, Wang Y, Li S, Chakravarty SD, Chan D, Shawi M, Yang YW, Thaҫi D, Rahman P. Long-Term Safety of Guselkumab in Patients with Psoriatic Disease: An Integrated Analysis of Eleven Phase II/III Clinical Studies in Psoriasis and Psoriatic Arthritis. Drug Saf. 2024 Jan;47(1):39-57. doi: 10.1007/s40264-023-01361-w. Epub 2023 Oct 31. PMID 37906417
- [Derived] Schett G, Chen W, Gao S, Chakravarty SD, Shawi M, Lavie F, Zimmermann M, Sharaf M, Coates LC, Siebert S. Effect of guselkumab on serum biomarkers in patients with active psoriatic arthritis and inadequate response to tumor necrosis factor inhibitors: results from the COSMOS phase 3b study. Arthritis Res Ther. 2023 Aug 16;25(1):150. doi: 10.1186/s13075-023-03125-4. PMID 37587493
- [Derived] Rahman P, Boehncke WH, Mease PJ, Gottlieb AB, McInnes IB, Shawi M, Wang Y, Sheng S, Kollmeier AP, Theander E, Yu J, Leibowitz E, Marrache AM, Coates LC. Safety of Guselkumab With and Without Prior Tumor Necrosis Factor Inhibitor Treatment: Pooled Results Across 4 Studies in Patients With Psoriatic Arthritis. J Rheumatol. 2023 Jun;50(6):769-780. doi: 10.3899/jrheum.220928. Epub 2023 Jan 15. PMID 36642439
- [Derived] Coates LC, Gossec L, Theander E, Bergmans P, Neuhold M, Karyekar CS, Shawi M, Noel W, Schett G, McInnes IB. Efficacy and safety of guselkumab in patients with active psoriatic arthritis who are inadequate responders to tumour necrosis factor inhibitors: results through one year of a phase IIIb, randomised, controlled study (COSMOS). Ann Rheum Dis. 2022 Mar;81(3):359-369. doi: 10.1136/annrheumdis-2021-220991. Epub 2021 Nov 24. PMID 34819273
- See also: Link to results on EudraCT registry. — https://www.clinicaltrialsregister.eu/ctr-search/trial/2018-003214-41/results